CLINICAL TRIAL: NCT03642301
Title: Dosing of Carcinogenic Complexes Such as Urinary O-toluidine and Hemoglobin Adducts From O-toluidine in Blood After Intrathecal Administration of 50 mg Hyperbaric Prilocaine
Brief Title: Dosing of Carcinogenic Complexes After Anesthesia With Intrathecal Hyperbaric Prilocaine.
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Collaborators: Ruhr University of Bochum (Other); Hôpital de Braine-l'Alleud (Other)
Responsible Party: Sponsor
Other Study IDs: B076201836443
Record Dates: First submitted 2018-07-24; First posted 2018-08-22 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Anesthesia
Keywords: Hemoglobin adducts from o-toluidine in blood; Urinary o-toluidine; Intrathecal anesthesia; Hyperbaric prilocaine; Ambulatory surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood (2 samples) and Urine (4 samples)
Oversight: Data Monitoring Committee: No

SUMMARY:
The prilocaine is a very common local anesthetic that has the disadvantage of being metabolized to o-toluidine, a human carcinogen.

Hyperbaric 2% prilocaine (HP), recently developped, is increasingly used for spinal anesthesia in ambulatory surgery. But the formation of carcinogenic metabolites induced by the hyperbaric prilocaine is not yet known. The aim of this study is to investigate whether the intrathecal administration of 50 mg hyperbaric prilocaine induces also the formation of carcinogenic complexes such as urinary o-toluidine and hemoglobin adducts from o-toluidine in blood.

ELIGIBILITY:
Inclusion Criteria:

* Age : > 18 years and < 80years
* American Society of Anesthesiology (ASA) score : I-II
* Height between 160cm and 180cm

Exclusion Criteria:

* Cardiac Disease (Aortic stenosis, heart failure...)
* coagulation disorder (International Normalized Ratio (INR) > 1.3; platelets <80 000/mm³)
* Allergic to local anesthetics
* Smoker

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient scheduled for an ambulatory surgery
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-03-27 (Actual)

PRIMARY OUTCOMES:
Hemoglobin adducts from o-toluidine in blood | Time 0 (before surgery)
  Hemoglobin adducts from o-toluidine in blood is measured before surgery (at admission)
Hemoglobin adducts from o-toluidine in blood | Time 24 hours after intrathecal prilocaine injection
  Hemoglobin adducts from o-toluidine in blood is measured at 24 hours after intrathecal prilocaine injection
Urinary o-toluidine | Time 0 (before surgery)
  Urinary o-toluidine is measured before surgery (at admission)
Urinary o-toluidine | Time 6 hours after intrathecal prilocaine injection
  Urinary o-toluidine is measured at 6 hours after intrathecal prilocaine injection
Urinary o-toluidine | Time 12 hours after intrathecal prilocaine injection
  Urinary o-toluidine is measured at 12 hours after intrathecal prilocaine injection
Urinary o-toluidine | Time 24 hours after intrathecal prilocaine injection
  Urinary o-toluidine is measured at 24 hours after intrathecal prilocaine injection

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Guntz, MD, Study Director — Université Libre de Bruxelles (ULB), Braine-l'Alleud Hospital; Panayota Kapessidou, MD,PhD, Principal Investigator — University Hospital Saint-Pierre (CHU Saint-Pierre), Université Libre de Bruxelles (ULB)
Locations (1):
- Braine-l'Alleud Hospital, Braine-l'Alleud, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaber K, Harreus UA, Matthias C, Kleinsasser NH, Richter E. Hemoglobin adducts of the human bladder carcinogen o-toluidine after treatment with the local anesthetic prilocaine. Toxicology. 2007 Jan 5;229(1-2):157-64. doi: 10.1016/j.tox.2006.10.012. Epub 2006 Oct 29. PMID 17129655
- [Background] Camponovo C, Fanelli A, Ghisi D, Cristina D, Fanelli G. A prospective, double-blinded, randomized, clinical trial comparing the efficacy of 40 mg and 60 mg hyperbaric 2% prilocaine versus 60 mg plain 2% prilocaine for intrathecal anesthesia in ambulatory surgery. Anesth Analg. 2010 Aug;111(2):568-72. doi: 10.1213/ANE.0b013e3181e30bb8. Epub 2010 Jun 7. PMID 20529983
- [Background] Guntz E, Latrech B, Tsiberidis C, Gouwy J, Kapessidou Y. ED50 and ED90 of intrathecal hyperbaric 2% prilocaine in ambulatory knee arthroscopy. Can J Anaesth. 2014 Sep;61(9):801-7. doi: 10.1007/s12630-014-0189-7. Epub 2014 Jun 7. PMID 24906303
- [Background] Gebhardt V, Herold A, Weiss C, Samakas A, Schmittner MD. Dosage finding for low-dose spinal anaesthesia using hyperbaric prilocaine in patients undergoing perianal outpatient surgery. Acta Anaesthesiol Scand. 2013 Feb;57(2):249-56. doi: 10.1111/aas.12031. Epub 2012 Nov 30. PMID 23199005
- [Background] Bohm F, Schmid D, Denzinger S, Wieland WF, Richter E. DNA adducts of ortho-toluidine in human bladder. Biomarkers. 2011 Mar;16(2):120-8. doi: 10.3109/1354750X.2010.534556. Epub 2010 Nov 30. PMID 21117897
- [Derived] Guntz E, Carini A, Koslitz S, Bruning T, Kapessidou P, Weiss T. Quantification of systemic o-toluidine after intrathecal administration of hyperbaric prilocaine in humans: a prospective cohort study. Arch Toxicol. 2021 Mar;95(3):925-934. doi: 10.1007/s00204-021-02973-w. Epub 2021 Jan 21. PMID 33475793